CLINICAL TRIAL: NCT02232711
Title: Evaluation of Accuracy and Ease of Use of the FilmArray™ Respiratory Panel (RP EZ) in a CLIA-Waived Clinical Setting
Status: Completed | Type: Observational
Sponsor: BioFire Diagnostics, LLC (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SDY-014162; HDTRA1-09-C0068 (Other Grant/Funding Number: Defense Threat Reduction Agency)
Record Dates: First submitted 2014-08-28; First posted 2014-09-05 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Upper Respiratory Infections
Keywords: multiplex, polymerase chain reaction, PCR, BioFire, respiratory infection, infectious disease, point of care, CLIA waived, rapid diagnostics
MeSH Terms: conditions — Respiratory Tract Infections; Pathologic Complete Response; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab (NPS) specimens
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the accuracy and ease-of-use of a simplified FilmArray Respiratory Panel test (FilmArray RP EZ) when performed according to the manufacturer's instructions by personnel in laboratories holding Clinical Laboratory Improvement Amendments (CLIA) waivers (or equivalent) on nasopharyngeal swab samples obtained from volunteers with signs and/or symptoms of a respiratory infection. The study data will be used to support an application to the FDA for CLIA-waived categorization of FilmArray RP EZ. It is hypothesized that the results of the FilmArray RP EZ test performed in a laboratory with CLIA waiver with be 95% accurate when compared to FilmArray RP testing performed in a lab with a moderate or high complexity CLIA certification.

ELIGIBILITY:
Inclusion Criteria:

* Displays signs and/or symptoms of respiratory infections
* Adult patients must provide informed consent
* Parental consent for children (<18)

Exclusion Criteria:

* Adult patients unable to provide informed consent
* Children that are currently in foster care, or are wards of the state

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with signs and/or symptoms of respiratory infections
Sampling Method: Non-Probability Sample
Enrollment: 1082 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of FilmArray RP EZ System in detecting cause of respiratory illness | 1.5 hour
  In general, performance of the FilmArray RP EZ test in the CLIA-waived setting is expected to meet at least 95% positive and negative percent agreement with the results obtained from FilmArray RP in the moderate/high- complexity setting for each pathogen on the panel.

SECONDARY OUTCOMES:
Epidemiology of respiratory infections in a CLIA-waived setting | Up to 9 months
  Seasonality and rate of respiratory infection at each of the CLIA-waived sites using the FilmArray RP EZ to collect prospectively enrolled specimens will be evaluated at the end of the study.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Naval Health Research Center, San Diego, California
  - Barnes-Jewish/Washington University School of Medicine, St Louis, Missouri
  - UTMB Primary Care Pavilion, Galveston, Texas
  - South Main Clinic, Salt Lake City, Utah

REFERENCES:
- [Background] Barenfanger J, Drake C, Leon N, Mueller T, Troutt T. Clinical and financial benefits of rapid detection of respiratory viruses: an outcomes study. J Clin Microbiol. 2000 Aug;38(8):2824-8. doi: 10.1128/JCM.38.8.2824-2828.2000. PMID 10921934
- [Background] Buller RS. Molecular detection of respiratory viruses. Clin Lab Med. 2013 Sep;33(3):439-60. doi: 10.1016/j.cll.2013.03.007. PMID 23931834
- [Background] Fairfax MR, Salimnia H. Diagnostic molecular microbiology: a 2013 snapshot. Clin Lab Med. 2013 Dec;33(4):787-803. doi: 10.1016/j.cll.2013.08.003. PMID 24267186